CLINICAL TRIAL: NCT06275100
Title: PREhabilitation in Patients Awaiting Acute Inpatient Cardiac SurgEry
Acronym: (PREP-ACE)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hull (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HUTH
Record Dates: First submitted 2023-10-16; First posted 2024-02-23 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Cardiac Disease; Aortic Valve Disease; Coronary Artery Disease; Endocarditis; Valve Heart Disease
MeSH Terms: conditions — Heart Diseases; Aortic Valve Disease; Coronary Artery Disease; Endocarditis; Heart Valve Diseases | interventions — Preoperative Exercise; Exercise

STUDY DESIGN:
Intervention Model Description: Single arm pilot feasibility study in acute inpatients waiting for cardiac surgery. Intervention is a prehabilitation program
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prehabilitation arm (Experimental): Participants will be exposed to physical and psychological prehabilitation whilst waiting for surgery. The prehabilitation will not alter the surgical waiting time or any medical intervention but aims to work around patient's essential care.
  Physical/ exercise component has a directly supervised component (aerobic exercise) and an unsupervised portion (Inspiratory muscle training and strength training) which is done via an app or leaflet depending on participant's preference. Participants will be given a guide number of exercises to do in their own time throughout the day.
  The psychological component consist of a psychoeducation booklet, meditation audio and signposting if they require further assistance. The psychoeducation component is voluntary.
  Interventions: Other: Prehabilitation

INTERVENTIONS:
Other: Prehabilitation — Participants will be exposed to exercise and psychoeducation. Aerobic exercise will be on a cycle ergometer tailored to their capability and will aim for a low to moderate intensity.The patients will be exercised using the intermittent protocol of alternating 1 minute moderate and 1 minute low intensity aerobic exercise. This duration can be gradually increased during subsequent sessions depending on the patient's ability. Aerobic exercise will be conducted 2- 3 times per week depending on patient's ability.
  In addition, participants are expected to do strength and inspiratory muscle training in their own time.
  The psychoeducation booklet and audio are designed with input from in-house clinical psychologist. The aim of the booklet is to explain the emotions they may feel whilst being in hospital, symptoms of anxiety, suggest how to manage anxiety, behavioural strategies that may help and signposting if they require further support.
  Other Names: exercise; psychological

SUMMARY:
This is a single centre, single arm pilot feasibility study to determine the feasibility and practicality of prehabilitation in acute inpatients waiting for cardiac surgery. We will be looking into participant eligibility, acceptability, recruitment rates, completion rates and barriers to implementing a prehabilitation programme. Secondary outcomes include safety (incidence of adverse events directly related to the study), improvement in 6 minutes walk test (6MWT), hand grip strength, quality of life, and spirometry. At the end of the trial, we will be seeking the feedback of the participants to help us improve the design further.

DETAILED DESCRIPTION:
Prehabilitation is a process of preparing a patient for major surgery with the aim of improving their outcome and recovery. Prehabilitation has shown benefits such as reduced post-operative complications and shorter inpatient stay in elective cardiac surgery population. There is currently no published research looking into the benefit of prehabilitation in acute inpatients.

I am currently doing an MD focusing on inpatients waiting for acute cardiac surgery in Castle Hill Hospital (CHH). The rationale for this is based on National Institute for Cardiovascular Outcomes Research (NICOR) report indicating that acute cardiac surgery waiting times increased, ranging from 7 to 24 days. Traditionally, inpatients are asked to have bed rest. However, this affects patient's mental and physical wellbeing, and hence negatively impact outcome.

The project consist of three parts. The first is an analysis of patients who had cardiac surgery in 2022 based on cardiac surgery audit data which is routinely collected for all patients. The purpose of this study is to assess the waiting times for acute cardiac surgery in East Yorkshire and describe the demographic and potential impact of the waiting times on these patients. We have sought local governance approval for this section as it involves data that is routinely collected in the department.

The second part of the project is a survey amongst patients waiting for acute cardiac surgery to gauge patient interest, how to engage them, opinion on design and potential problems that needs to be addressed.

The third and main part of the project is a single centre, single arm, prospective, pilot feasibility trial aiming to recruit 20 acute inpatients. The primary objective of the trial is to investigate the feasibility, acceptability and completion rates of prehabilitation. The secondary objective is to identify any potential improvement and safety concerns. The intervention involves exercise and anxiety management. The interventions will start as soon as the patient is recruited, end on the day before surgery and not impact the date of their surgery.

We have received ethical approval from Hull York Medical School (HYMS) ethics committee for the second and third part of the project. In addition to this, we have also applied for Research Ethics Committee (REC) approval in Integrated Research Application System (IRAS). We are awaiting the REC approval.

ELIGIBILITY:
Inclusion Criteria:

* All patients over the age of 18 scheduled for acute cardiac surgery in CHH will be given consideration to participate in this clinical trial.

Exclusion Criteria:

* Patients who are unable or unwilling to participate in any of the elements of prehabilitation will be excluded. These include those that have cognitive disability (including unconsciousness), cardiac or clinical instability, functional or anatomical impairment which impairs ability to participate, language barrier or patient refusal. Patients that have impending surgery within 72 hours of arrival to hospital will be excluded. Patients who are awaiting surgery in district hospitals or outside of Castle Hill Hospital will be excluded. A non-exhaustive list of exclusion criteria is included below.

Cardiac/ clinical instability such as:

* Recurrent unstable angina/ crescendo angina
* Untreated decompensated heart failure
* Malignant arrhythmias awaiting treatment
* Resting tachycardia (HR>100 bpm)
* Left ventricular outflow obstruction such as Aortic Stenosis with pre-syncopal or syncopal symptoms
* Unresolved acute pericarditis or myocarditis
* Second or third degree heart block without pacemaker
* Aortic Dissection
* Myxoma

Functional/ anatomical impairment such as:

* Severe musculoskeletal conditions that would prohibit exercise
* Amputees
* Registered blind

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-04-03 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Feasibility of prehabilitation in acute inpatients waiting for cardiac surgery | We estimate from patient recruitment to day before surgery can be between 7 days and 4 weeks. Intervention will start as soon as patient is recruited and end the day before their surgery
  We will be assessing the eligibility, recruitment rate, deliverability, logistical, practicality, completion rate, achievability and acceptability of the program. This is based on the recruitment as well as participant feedback interview.

SECONDARY OUTCOMES:
Efficacy of prehabilitation | Assessment will be done on day 0 (recruitment), day 7 and day 14 or day before surgery
  To identify a signal of efficacy for positive changes in physical health exercise, mental wellbeing and quality of life. This is done by assessing participants changes in 6 minutes walk test (6MWT).
Efficacy of prehabilitation | Assessment will be done on day 0 (recruitment), day 7 and day 14 or day before surgery
  To identify a signal of efficacy for positive changes in physical health exercise, mental wellbeing and quality of life. This is done by assessing participants changes in hand grip strength.
Efficacy of prehabilitation | Assessment will be done on day 0 (recruitment), day 7 and day 14 or day before surgery
  To identify a signal of efficacy for positive changes in physical health exercise, mental wellbeing and quality of life. This is done by assessing participants changes in EuroQol questionnaire (EQ5D5L).
Efficacy of prehabilitation | Assessment will be done on day 0 (recruitment), day 7 and day 14 or day before surgery
  To identify a signal of efficacy for positive changes in physical health exercise, mental wellbeing and quality of life. This is done by assessing participants changes in Cardiac Anxiety Questionnaire (CAQ).
Efficacy of prehabilitation | Assessment will be done on day 0 (recruitment), day 7 and day 14 or day before surgery
  To identify a signal of efficacy for positive changes in physical health exercise, mental wellbeing and quality of life. This is done by assessing participants changes in spirometry.
Complication rate | Day 0 (pre op) to day of patient discharge or 30 post op
  To identify differences in length of hospital stay, complications and readmission rates to hospital following surgery compared to usual care. This is done by comparing our outcomes with the hospital's standard care. Outcome from standard care will be obtained from hospital audit data
Safety of Prehabilitation in acute inpatients waiting for surgery | day 0 to day before surgery
  Throughout the study, we will be collecting information on adverse events, complications which may or may not be related to the intervention(s)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Raut, Principal Investigator — University of Hull
Locations (1):
- Hull University Teaching Hospital, Hull, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No personal data will be shared. However, if requested, anonymised data pertaining to the study can be shared

REFERENCES:
- [Derived] Raut S, Hales A, Twiddy M, Dixon L, Ngaage D, Yates D, Danjoux G, Ingle L. Multimodal prehabilitation in people awaiting acute inpatient cardiac surgery: Study protocol for a pilot feasibility trial (PreP-ACe). PLoS One. 2025 Mar 10;20(3):e0307341. doi: 10.1371/journal.pone.0307341. eCollection 2025. PMID 40063583

DOCUMENTS (2):
  • Study Protocol (2023-11-06): https://cdn.clinicaltrials.gov/large-docs/00/NCT06275100/Prot_000.pdf
  • Informed Consent Form (2023-11-06): https://cdn.clinicaltrials.gov/large-docs/00/NCT06275100/ICF_001.pdf